CLINICAL TRIAL: NCT05976854
Title: Effects of an Online Intervention Based on Pain Neuroscience Education for Women with Pregnancy-related Lumbopelvic Pain
Brief Title: Online Intervention Based on Pain Neuroscience Education for Women with Pregnancy-related Lumbopelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-65
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Prenatal Education

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain neuroscience education (PNE) (Experimental): The patients in the intervention group will receive, in addition to the prenatal educational content, the 12 PNE lessons in audiovisual format. Each lesson will last between 10-15 minutes. The contents of PNE will be an adaptation, focused on the context of a pregnant woman, of the Butler & Moseley postulates. These contents have already been previously adapted according to the nature of the patients' pain, both in chronic pain and in acute pain. In summary, the participants will receive a detailed explanation about the biopsychosocial component of pain through the use of diagrams, metaphors and practical examples. In turn, the objectives of this program could be summarized as: (1) Reformulate erroneous beliefs about pain, (2) Inform about the biology and protective nature of pain and (3) Provide techniques to reduce kinesiophobia and, consequently, promote physical activity, with the beneficial effect it entails for patients with pain.
  Interventions: Other: Pain neuroscience education; Other: Prenatal education
- Prenatal education (PE) (Other): Patients assigned to the PE group will receive different content on standard PE based on the Pregnancy and Postpartum Clinical Practice Guide, consisting of general information about pregnancy (visits and monitoring of pregnancy, diet, phases of delivery, lactation, etc.), as well as specific recommendations for lumbopelvic pain associated with pregnancy. These contents will be developed by midwives from the participating hospitals. Participants will receive 12 educational sessions, with an estimated duration of 10 minutes each.
  Interventions: Other: Prenatal education

INTERVENTIONS:
Other: Pain neuroscience education — The patients in the intervention group will receive, in addition to the prenatal educational content, the 12 Pain neuroscience education lessons in audiovisual format. Each lesson will last between 10-15 minutes. The contents of PNE will be an adaptation, focused on the context of a pregnant woman, of the Butler & Moseley postulates. These contents have already been previously adapted according to the nature of the patients' pain, both in chronic pain and in acute pain. In summary, the participants will receive a detailed explanation about the biopsychosocial component of pain through the use of diagrams, metaphors and practical examples. In turn, the objectives of this program could be summarized as: (1) Reformulate erroneous beliefs about pain, (2) Inform about the biology and protective nature of pain and (3) Provide techniques to reduce kinesiophobia and, consequently, promote physical activity, with the beneficial effect it entails for patients with pain.
  Arms: Pain neuroscience education (PNE)
Other: Prenatal education — The standard prenatal education is based on the Pregnancy and Postpartum Clinical Practice Guide, consisting of general information about pregnancy (visits and monitoring of pregnancy, diet, phases of delivery, lactation, etc.), as well as specific recommendations for lumbopelvic pain associated with pregnancy. These contents will be developed by midwives from the participating hospitals. Participants will receive 12 educational sessions, with an estimated duration of 10 minutes each.

SUMMARY:
60-70% of pregnant women suffer from pregnancy-related lumbopelvic pain. In the general population, patient education is the first line of treatment. For pregnant women with LBP, the guidelines are the same as for the general population. In fact, prenatal education programs specifically collect recommendations and educational strategies for managing this pain. Within educational strategies, education in the neuroscience of pain has gained special relevance in recent years due to its positive results in reducing pain in patients with low back pain. Despite the beneficial effects shown in patients with low back pain, its use has not yet been explored, to our knowledge, in women with pregnancy-related lumbopelvic pain.

DETAILED DESCRIPTION:
60-70% of pregnant women suffer from pregnancy-related lumbopelvic pain. Its multifactorial origin makes it difficult to establish an appropriate treatment for pain control. In the general population, patient education is the first line of treatment. For pregnant women with LBP, the guidelines are the same as for the general population. In fact, prenatal education programs specifically collect recommendations and educational strategies for managing this pain. Within educational strategies, education in the neuroscience of pain has gained special relevance in recent years due to its positive results in reducing pain in patients with low back pain. This type of education is based on reconceptualizing pain through teaching the neurobiological mechanisms that underlie the pain experience. Despite the beneficial effects shown in patients with low back pain, its use has not yet been explored, to our knowledge, in pregnant women with pregnancy-related low back and pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women older than 18 years, who are in the early third trimester of pregnancy;
* minimum score of 3/10 on the numerical pain scale over the past week.

Exclusion Criteria:

* multiple pregnancy;
* previous spinal surgery;
* presence of psychiatric disorders;
* women who have participated in similar programs or interventions before enrollment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  The primary outcome will be mean pain intensity over the previous week assessed using an 11-point numerical rating scale (range, 0 [no pain] to 10 [worst pain imaginable]).

SECONDARY OUTCOMES:
Disability | 4 weeks
  The Roland Morris questionnaire will be used. This is a validated questionnaire for the Spanish population and has previously been used in women with lumbopelvic pain. The questionnaire assesses the degree of physical disability in patients with non-specific low back pain and is made up of 24 items that describe daily activities that may be difficult to perform due to low back pain. A point is added to each item marked "yes", and a maximum score of 24 points can be obtained. The greater the number of positive responses, the greater the disability.
Kinesiophobia | 4 weeks
  The short version of the Tampa TSK-11 kinesiophobia scale will be used The Spanish version of this scale has been validated in patients with acute and chronic low back pain. The scale consists of 11 items, in which each item receives a score from 1 to 4 on the Likert scale (1=strongly disagree; 4=strongly agree). The score ranges from 11 to 44 points, with higher scores indicating a greater fear of movement.
Pain catastrophizing | 4 weeks
  The pain catastrophizing scale is an instrument made up of 13 items (each item scores between 0 and 4), which measures the degree to which patients develop feelings and thoughts related to their nociceptive experience. This scale, which has a validated version for Spanish, shows adequate internal consistency.
Anxiety and depression | 4 weeks
  The Hospital Anxiety and Depression Scale (HADS) questionnaire will be used. This consists of 14 questions, of which 7 assess symptoms of anxiety (HADS-A) and 7 measure symptoms of depression (HADS-D). Each item scores from 0 to 3, with a score range in each subscale from 0-21. Scores of 0-7 indicate no anxiety or depression; scores between 8-10 indicate medium levels; scores of 11-14 indicate moderate levels and scores of 15-21 indicate severe levels of anxiety or depression. The HADS scale has good internal consistency, reliability, and validity.
Level of physical activity | 4 weeks
  The abbreviated version of the international physical activity questionnaire (International Physical Activity Questionnaire - IPAQ - short) will be used. This is a self-administered questionnaire consisting of 7 items and collecting information on physical activity performed in the last 7 days. This questionnaire has been previously validated in 12 countries and shows adequate psychometric properties. The short version (IPAD-SF) has shown acceptable validity in the Spanish adult population.

CONTACTS AND LOCATIONS:
Locations (1):
- JF Lisón, Alfara del Patriarca, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia-Lucas C, Chen E, Serrano-Raya L, Boldo-Roda A, Arguisuelas MD, Suso-Marti L, Pardo J, Amer-Cuenca JJ, Lison JF, Bivia-Roig G. Association between lumbopelvic pain in pregnancy and fear of childbirth: a multicenter cross-sectional case-control study. BMC Pregnancy Childbirth. 2025 Nov 17;25(1):1215. doi: 10.1186/s12884-025-08425-y. PMID 41250063